CLINICAL TRIAL: NCT03204825
Title: Pain Management and Patient Education for Physical Activity in Intermittent Claudication (PrEPAID): Feasibility Randomised Controlled Trial
Brief Title: Pain Management and Patient Education for Physical Activity in Intermittent Claudication (PrEPAID)
Acronym: PrEPAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); University of Glasgow (Other); Northumbria University (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16 044
Record Dates: First submitted 2017-04-25; First posted 2017-07-02 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: Patient education; Pain management; Transcutaneous electrical nerve stimulation; Physical activity; Feasibility
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Agnosia; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation; Educational Status

STUDY DESIGN:
Intervention Model Description: 2x2 randomised feasibility controlled trial blinded for primary outcome
Who Masked: Participant, Outcomes Assessor
Masking Description: Primary outcome assessors will be blinded for patient group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active TENS (Experimental): Participants in the TENS groups will be provided with a TENS machine and training at the baseline visit to the Clinical research Facility (CRF). They will be instructed to use it daily as their symptoms require for 6 weeks. The active group will receive High Frequency-TENS (120 Hz, 200µs and a patient-determined intensity of ''strong but comfortable'').
  Interventions: Device: Active TENS
- Placebo TENS (Placebo Comparator): Placebo TENS : Participants will receive the same model, programmed settings and instructions for use as those in the active group except that the device will be set to an ineffective stimulation (120 Hz, 200µs and a patient-determined intensity of '6mA). For the purpose of blinding, participants will be told that different dosages of TENS are being tested, some of which where the stimulation might not be perceivable even though the device is working.
  Interventions: Device: Placebo TENS
- Patient-Centred Education (Experimental): Patient-Centred Education : a one-off three-hour workshop of structured group education (4-5 persons in each group) and three 2-weekly phone calls. The aim will be to modify patients' illness beliefs and perceptions about IC/PAD by educating them on disease pathology and management philosophy. After the workshop, each patient will be supported to set goals for walking, develop an action plan regarding how these goals will be met and encouraged to repeat this process for each new walking goal.
  Interventions: Behavioral: Patient-Centred Education
- Patient-Centred Education + Active TENS (Experimental): Combination of Patient-Centred Education arm and Active TENS arm.
  Interventions: Device: Active TENS; Behavioral: Patient-Centred Education

INTERVENTIONS:
Device: Active TENS — TENS is a form of electrical stimulation that provides symptomatic pain relief that is used extensively within the health-care setting. It is a non-invasive modality; packaged in a small, portable unit that is easy to apply via small electrodes placed on the skin.
  Other Names: TENS; TNS; Transcutaneous Nerve Stimulation; Transcutaneous Electrical Nerve Stimulation
  Arms: Active TENS; Patient-Centred Education + Active TENS
Behavioral: Patient-Centred Education — Group education for patients with peripheral arterial disease and intermittent claudication about their condition, improving patient ownership, and promoting self-managed walking
  Other Names: Education; SEDRIC; Structured patient-centred education intervention
  Arms: Patient-Centred Education; Patient-Centred Education + Active TENS
Device: Placebo TENS — TENS device use with setting so that the stimulation delivered is ineffective
  Other Names: P-TENS; Placebo Transcutaneous Electrical Nerve Stimulation
  Arms: Placebo TENS

SUMMARY:
Peripheral Arterial disease is a common condition which causes narrowing of the arteries. The most common symptom that patients with PAD experience is Intermittent Claudication (IC), pain in the lower limb(s) on exertion, which is relieved by rest. IC reduces patients' quality of life (QoL) by limiting their ability to walk and engage in daily activities. Regular exercise and physical activity (PA) are central to the management of PAD and help to improve walking distances and reduce the risks associated with PAD such as heart attack and stroke. However, exercise and PA in this population is often limited due to pain. Investigators have shown that Transcutaneous Electrical Nerve Stimulation (TENS) can help to reduce pain and increase walking distance in patients with PAD. Investigators have also shown that educating patients about their condition and helping them to set goals has the potential to increase PA, and quality of life. This study will examine the feasibility of designing a definitive trial that investigates whether TENS can improve the physical activity of patients with PAD when delivered alone and/or alongside a patient education programme.

DETAILED DESCRIPTION:
Peripheral Arterial disease (PAD) affects 2.7 million people in the United Kingdom (UK). The most common symptom that patients experience is Intermittent Claudication (IC), which is pain in the buttock, calf or thigh precipitated by exercise and relieved by rest. The underlying cause of PAD is atherosclerosis, which leads to arterial stenosis, inadequate blood flow and build-up of lactic acid during exercise. Patients with IC have impaired quality of life due to reduced physical capacity. Furthermore, due to the diffuse nature of atherosclerosis and the involvement of other arterial beds, they have 3-4 times increased mortality compared to age and sex matched controls.

Patients with symptomatic PAD should receive the same secondary prevention management as patients with symptomatic coronary artery disease. Improving daily physical activity (PA) is particularly important in individuals with IC as lower PA levels have been recognised as a strong predictor of increased morbidity and mortality in this population. Current National Institute for Health and Care Excellence (NICE) guidelines recommend the use of supervised exercise programmes (SEPs), encouraging patients "to exercise to the point of maximal pain", as first line treatment. SEPs has been shown to be cost-effective when compared to other treatment options such as endovascular intervention and surgical revascularisation. However, while systematic reviews show that SEPs lead to a significant improvement in the absolute walking distances of patients with IC on a treadmill, it is unclear if this is sustained or leads to improvement in daily PA. Furthermore, due to the considerable extra resources required to deliver the recommended 3 months exercise programme (30-45 minutes 3x weekly), SEPs are not always routinely available to National Health Service (NHS) patients, and time and travel costs tend to lead to low patient uptake and high attrition rates. Therefore, investigating the feasibility of using low-cost, patient-centred interventions that can support increased PA is warranted.

Lack of self-efficacy, attributed to poor understanding of the disease and uncertainty regarding the importance of exercise, has been shown to be a major barrier to exercise uptake in this population. Educating patients with IC about their disease pathology and the benefits of walking is key to enhancing success of secondary prevention strategies for people with IC. Investigators recently piloted a structured, patient-centred education intervention (SEDRIC) with the specific aim of educating patients with IC about their condition, improving patient ownership, and promoting self-managed walking. In addition to improved treadmill walking distances, investigators found out that there was a trend for patients to increase their daily PA.

For patients with IC to gain benefits of secondary prevention, exercising beyond the point when pain occurs is recommended, representing another barrier to engagement in PA. Despite this, investigators' systematic review found that pain management as a route to facilitate exercise and PA has rarely been explored. Recent interest has focused on the use of TENS (a low-cost, non-invasive pain management device) to improve angiogenesis, muscle function, pain and walking distances in patients with IC. TENS has a strong placebo effect in pain conditions, and testing effectiveness against placebo is advocated. In a proof-of-concept pilot study, Investigators demonstrated that TENS could significantly improve pain and increase treadmill walking distances above placebo levels. Our exploratory study also established that home use of TENS was both acceptable and provided self-reported improvement in PA in individuals with IC.

Although patient-centred education (SEDRIC) and TENS have both demonstrated potential to improve daily PA in people with IC, the use of these components in combination has not previously been evaluated. Investigators therefore propose a 2 x 2 (TENS versus placebo TENS x SEDRIC versus no additional education) feasibility Randomised Controlled Trial (RCT) that will compare use of TENS against placebo TENS with and without a patient-centred education programme.

Investigators have conducted a series of pilot studies underpinning both aspects of the intervention. Investigators have demonstrated in an experimental lower limb ischaemic pain model in healthy volunteers (n=28) that TENS significantly reduced onset of pain (by 29 seconds; 23%), tolerance of pain (by 203 seconds; 53%) and the pain endurance (by 173 seconds; 67%), compared to placebo TENS. Following this, in a proof-of-concept pilot study, investigators demonstrated that TENS when applied to patient with IC exercising on a treadmill (n=40) significantly improved absolute claudication distance (ACD) above placebo levels (approx. mean individual increase in ACD of 40%, p=.025, r= .53). Our phase 2 study also established that home use of TENS was both acceptable and provided self-reported improvement in PA in individuals with IC. Investigators have not assessed the ability of TENS to improve ACD when used during daily life.

Similarly, this research group developed and piloted SEDRIC, a structured, patient-centred education intervention with the specific aim of educating patients about their condition, improving patient ownership, and promoting self-managed walking. Investigators found that in patients with PAD (n=14), treadmill walking distances (30%) and quality of life (32%) improved from baseline after 6 weeks of structured education, and there was a trend for patients to increase their daily PA (approx. 8% change from baseline).

The aim is to determine the feasibility of electrical stimulation via a low-cost CE-marked device used within a patient centred education programme to improve walking distances in patients with PAD.

The following research questions will be answered by this project:

1. What is the feasibility (i.e. recruitment and retention rates, adherence, safety, sample size for a definitive trial, potential for effectiveness) of conducting a definitive RCT comparing TENS with and without patient-centred education?
2. How acceptable are TENS and patient-centred education as interventions on their own or in combination in patients with IC?

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of symptomatic Peripheral Arterial Disease (PAD) including resting Ankle Brachial Pressure Index (ABPI) <0.9 in at least one leg
* Stable IC for ≥3 months
* Walking limited primarily by claudication
* Able to exercise on a treadmill
* Able to read and speak English to a level allowing satisfactory completion of the study procedures
* Able to provide written informed consent for participation

Exclusion Criteria:

* Planned surgical or endovascular intervention for PAD within the next 3 months
* Critical limb ischaemia
* The presence of any absolute contraindications to exercise testing/training as defined by the American College of Sports Medicine (ACSM)
* Previous experience of using TENS/ structured patient education for PAD
* Contraindications to TENS (including epilepsy, dermatological conditions, indwelling electrical pumps/pacemakers) and inability to apply TENS independently.
* Patients who require walking aids including artificial limbs
* Major surgery, myocardial infarction or stroke/ Transient Ischaemic Attack (TIA) in the previous 6 months
* Co-morbidities that cause pain or limit walking to a greater extent than IC (e.g. severe arthritis)
* >20% variation in baseline ACD on treadmill
* Severe peripheral neuropathies above the ankle.
* Participation in another research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Seenan, PT, PhD, Study Director — Glasgow Caledonian University; UKACHUKWU ABARAOGU, MSc, PT, Principal Investigator — Glasgow Caledonian University; Julie Brittenden, MD, FRCS, Study Chair — Queen Elizabeth University Hospital/University of Glasgow
Locations (1):
- Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow, Strathcylde, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abaraogu UO, Dall PM, Seenan CA. Patient education interventions to improve physical activity in patients with intermittent claudication: a protocol for a systematic mixed-studies review. BMJ Open. 2016 May 20;6(5):e011405. doi: 10.1136/bmjopen-2016-011405. PMID 27207628
- [Background] Tew GA, Humphreys L, Crank H, Hewitt C, Nawaz S, Al-Jundi W, Trender H, Michaels J, Gorely T. The development and pilot randomised controlled trial of a group education programme for promoting walking in people with intermittent claudication. Vasc Med. 2015 Aug;20(4):348-57. doi: 10.1177/1358863X15577857. Epub 2015 Apr 9. PMID 25858012
- [Background] Abaraogu UO, Ezenwankwo EF, Dall PM, Seenan CA. Living a burdensome and demanding life: A qualitative systematic review of the patients experiences of peripheral arterial disease. PLoS One. 2018 Nov 15;13(11):e0207456. doi: 10.1371/journal.pone.0207456. eCollection 2018. PMID 30440040
- [Background] Abaraogu U, Ezenwankwo E, Dall P, Tew G, Stuart W, Brittenden J, Seenan C. Barriers and enablers to walking in individuals with intermittent claudication: A systematic review to conceptualize a relevant and patient-centered program. PLoS One. 2018 Jul 26;13(7):e0201095. doi: 10.1371/journal.pone.0201095. eCollection 2018. PMID 30048501
- [Background] Abaraogu UO, Dall PM, Seenan CA. The Effect of Structured Patient Education on Physical Activity in Patients with Peripheral Arterial Disease and Intermittent Claudication: A Systematic Review. Eur J Vasc Endovasc Surg. 2017 Jul;54(1):58-68. doi: 10.1016/j.ejvs.2017.04.003. Epub 2017 May 18. PMID 28528678
- [Derived] Seenan C, Abaraogu U, Dall PM, Gilmour L, Tew G, Stuart W, Elders A, Brittenden J. Pain management and patient education interventions to increase physical activity in people with intermittent claudication (PrEPAID): a feasibility randomised controlled trial in the UK. BMJ Open. 2025 Jul 22;15(7):e105563. doi: 10.1136/bmjopen-2025-105563. PMID 40701603
- [Derived] Abaraogu UO, Dall PM, Brittenden J, Stuart W, Tew GA, Godwin J, Seenan CA. Efficacy and Feasibility of Pain management and Patient Education for Physical Activity in Intermittent claudication (PrEPAID): protocol for a randomised controlled trial. Trials. 2019 Apr 16;20(1):222. doi: 10.1186/s13063-019-3307-6. PMID 30992033

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was open for recruitment between August 2017 and March 2020. In total, 1030 people were screened for eligibility; 763 (74%) were ineligible, mainly because they were on the clinic lists due to other conditions e.g., Abdominal Aortic Aneurysm or venous disease (n=343, 45% of ineligible total) or had Critical Limb Ischaemia (CLI) (n=122, 16%). There were 172 individuals that either did not consent to participate or did not respond to invitation.
Pre-assignment Details: Participants underwent additional screening prior to randomisation in adherence with the inclusion criteria in the protocol. Thirty-nine participants did not pass screening, 38 (97%) due to having a greater than 20% variance in ACD between the first and second screening visits (one week apart). The other participant who did not pass screening was unable to walk on the treadmill.
Groups:
- Patient-Centred Education and Placebo TENS: Patient-Centred Education : a one-off three-hour workshop of structured group education (4-5 persons in each group) and three 2-weekly phone calls. The aim will be to modify patients' illness beliefs and perceptions about IC/PAD by educating them on disease pathology and management philosophy. After the workshop, each patient will be supported to set goals for walking, develop an action plan regarding how these goals will be met and encouraged to repeat this process for each new walking goal.
  Patient-Centred Education: Group education for patients with peripheral arterial disease and intermittent claudication about their condition, improving patient ownership, and promoting self-managed walking
  Placebo TENS : Participants will receive the same model, programmed settings and instructions for use as those in the active group except that the device will be set to an ineffective stimulation (120 Hz, 200µs and a patient-determined intensity of '6mA). For the purpose of blinding, participants will be told that different dosages of TENS are being tested, some of which where the stimulation might not be perceivable even though the device is working.
  Placebo TENS: TENS device use with setting so that the stimulation delivered is ineffective.
Period: Overall Study
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Started | 14 | 14 | 14 | 14
End of Intervention | 12 | 11 | 13 | 13
Completed | 13 | 10 | 12 | 10
Not Completed | 1 | 4 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education | Patient-Centred Education + Active TENS | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (9.7) | 69.1 (10.1) | 64.0 (5.5) | 66.9 (8.3) | 66.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 5 | 14
  Male | 10 | 13 | 10 | 9 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14 | 14 | 14 | 14 | 56
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (4.7) | 27.9 (3.9) | 30.2 (5.5) | 29.4 (4.3) | 28.5 (4.8)
Ankle Brachial Pressure Index [Mean (Standard Deviation); unit: Ratio of systolic BP - UL / LL] | 0.70 (0.21) | 0.74 (0.28) | 0.67 (0.15) | 0.66 (0.14) | 0.69 (0.20)
Initial Claudication Distance (ICD) [Mean (Standard Deviation); unit: Metres] | 84.4 (78.2) | 126.1 (165.2) | 130.2 (129.6) | 111.7 (162.3) | 113.1 (135.7)
Absolute Claudication Distance (ACD) [Mean (Standard Deviation); unit: Metres] | 243.7 (240.5) | 251.3 (266.5) | 370.9 (285.3) | 318.4 (321.6) | 296.1 (277.3)
Average daily number of steps ('000s) [Mean (Standard Deviation); unit: Steps per day] | 7.5 (7.1) | 4.9 (2.1) | 6.0 (2.8) | 5.1 (3.9) | 5.9 (4.4)
Average daily number of upright events [Mean (Standard Deviation); unit: Count] | 7.0 (2.9) | 6.1 (2.7) | 6.6 (2.9) | 6.1 (1.8) | 6.4 (2.5)
Average daily number of walking events [Mean (Standard Deviation); unit: Count] | 50.0 (24.0) | 50.2 (21.2) | 53.6 (26.0) | 46.4 (19.1) | 50.0 (22.2)
Event-based Claudication Index [Mean (Standard Deviation); unit: Ratio] | 7.3 (2.8) | 8.9 (4.4) | 8.4 (4.3) | 8.5 (6.3) | 8.3 (4.6)
SF-36 Physical Component Score [Mean (Standard Deviation); unit: units on a scale] — 36-Item Short Form Survey (SF-36). Self-completed by participants The physical component score (PCS) on the Short Form 36 (SF-36) health survey is a summary score that combines the first four domains of the survey: physical function, physical role, bodily pain, and vitality.
  The SF-36 is a 36-question survey that measures health across eight domains. Each domain is scored from 0 to 100, with higher scores indicating better health.
  units on a scale | 34.4 (7.5) | 32.5 (8.9) | 37.3 (5.2) | 38.1 (6.0) | 35.6 (7.2)
SF-36 Mental Component Score [Mean (Standard Deviation); unit: units on a scale] — 36-Item Short Form Survey (SF-36). Self-completed by participants
  The SF-36 is a self-report survey that assesses physical and mental health across eight domains:
  To calculate the MCS, you first calculate a raw score for each of the four mental health domains (Emotional role functioning, Social role functioning Mental health or emotional wellbeing, Vitality), then convert the raw score to a scale score. Scale is scored from 0-100 with higher scores representing greater quality of life.
  units on a scale | 23.9 (11.3) | 22.7 (11.7) | 25.3 (12.7) | 24.6 (13.9) | 24.1 (12.2)
Intermittent Claudication Questionnaire [Mean (Standard Deviation); unit: units on a scale] | 53.1 (16.0) | 53.2 (15.7) | 52.2 (15.4) | 47.6 (16.0) | 51.5 (15.5)
Geriatric Depression Scale (short-form) [Mean (Standard Deviation); unit: units on a scale] | 6.6 (4.2) | 5.1 (3.9) | 7.1 (4.6) | 6.4 (4.7) | 6.3 (4.3)
McGill Pain Questionnaire [Mean (Standard Deviation); unit: units on a scale] | 30.6 (13.6) | 22.2 (13.1) | 31.2 (14.4) | 29.4 (10.6) | 28.4 (13.1)
Pain Self-Efficacy Questionnaire [Mean (Standard Deviation); unit: units on a scale] | 35.8 (13.7) | 42.4 (14.3) | 36.5 (14.8) | 35.2 (13.9) | 37.5 (14.1)
Pain intensity (visual analogue scale) [Mean (Standard Deviation); unit: units on a scale] | 6.3 (2.3) | 6.2 (2.8) | 6.6 (2.4) | 5.5 (2.6) | 6.2 (2.5)
Brief Illness Perception Questionnaire [Mean (Standard Deviation); unit: units on a scale] | 47.2 (11.9) | 43.4 (10.1) | 49.8 (9.7) | 49.3 (10.4) | 47.4 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Absolute Claudication Distance (ACD) in Meters From Baseline
Description: Maximal walking distance on graded treadmill test
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: metres
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 12 | 11 | 13 | 13
metres
  Change scores from baseline to end of intervention (6 weeks) | -16.8 [-62.1 to 28.4] | -6.7 [-33.8 to 20.5] | 76.2 [17.0 to 135.4] | -0.9 [-44.2 to 42.4]
  Change scores from baseline to follow-up (18 weeks) | 25.0 [-26.8 to 76.7] | -17.6 [-41.0 to 5.8] | 89.2 [21.3 to 157.1] | -15.1 [-64.1 to 33.9]

2. Primary Outcome: Recruitment Rates
Description: Measure recruitment rates (ratio of patients who consent to participate to potentially eligible patient recorded via the study screening log
Time Frame: Recruitment
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: Eligible patients as identified by screening clinic lists.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 267
Participants | 95

3. Primary Outcome: Participant Retention Rate
Description: Ratio of patients who completed the intervention and outcome assessment to the patient who consented
Time Frame: End of study (18 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
Participants | 13 | 10 | 12 | 10

4. Primary Outcome: Adverse Events
Description: Record defined adverse events in all groups
Time Frame: End of study (18 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Patient-Centred Education + Active TENS | Active TENS | Patient-Centred Education and Placebo TENS | Placebo TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
Participants | 1 | 0 | 0 | 0

5. Primary Outcome: Uptake of Interventions
Description: Measure uptake of intervention via log of TENS use and attendance at education session and follow up phone calls
Time Frame: End of study (18 weeks)
Population: Population described as a whole rather than per-arm as data per arm was not recorded due to blinding. All participants were randomised to receive some type of TENS hence 56 total and 50% of participants received education, hence n=28.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Randomised to Receive TENS: Participants randomised to receive TENS.
- Attendance at Education Sessions.: Participants randomised to receive education.
- Attendance at Phone Call Follow-up: Participants randomised to education
Arm/Group | Participants Randomised to Receive TENS | Attendance at Education Sessions. | Attendance at Phone Call Follow-up
Number analyzed (Participants) | 56 | 28 | 28
Participants | 39 | 27 | 18

6. Secondary Outcome: Change in Initial Claudication Distance (ICD) in Meters From Baseline
Description: Onset distance of claudication pain on graded treadmill test
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: metres
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
metres
  Change from baseline to end of intervention (6 weeks) | 37.8 [5.9 to 69.8] | 23.2 [-17.0 to 163.5] | 107.6 [37.3 to 178.0] | 52.2 [5.0 to 99.4]
  Change from baseline to follow-up (18 weeks) | 55.2 [-11.4 to 121.7] | 77.1 [-83.4 to 237.5] | 122.7 [26.6 to 218.9] | 54.1 [-3.9 to 112.1]

7. Secondary Outcome: Change in Daily Number of Steps
Description: Change in daily number of steps (activpal step counts)
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: steps
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
steps
  Change from baseline to end of intervention (6 weeks) | -1568 [-3766 to 631] | -237 [-874 to 399] | 1076 [-758 to 2910] | 442 [-430 to 1314]
  Change from baseline to follow-up (18 weeks) | -1942 [-3239 to -646] | -183 [-1048 to 683] | 1615 [-2425 to 5654] | -1637 [-4010 to 736]

8. Secondary Outcome: Change in Total Number of Upright Events Per Day
Description: Total number of upright events per day (activpal upright even count)
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: upright events per day
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
upright events per day
  Change from baseline to end of intervention (6 weeks) | -1.1 [-8.6 to 6.3] | -2.3 [-6.9 to 2.4] | -3.9 [-13.5 to 5.6] | 1.7 [-2.3 to 5.7]
  Change from baseline to follow-up (18 weeks) | -2.1 [-8.4 to 4.1] | 2.5 [-3.8 to 8.9] | -4.7 [-9.2 to -0.2] | -3.4 [-13.0 to 6.1]

9. Secondary Outcome: Change in Total Number of Walking Events Per Day
Description: Total number of walking events per day (activpal walking event counts)
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: events per day
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
events per day
  Change from baseline to end of intervention (6 weeks) | -27.7 [-88.4 to 33.0] | -22.1 [-65.3 to 21.1] | -27.6 [-106.1 to 50.8] | 16.3 [-46.1 to 78.6]
  Change from baseline to follow-up (18 weeks) | -53.5 [-99.6 to -7.4] | 0.1 [-75.8 to 76.1] | -36.9 [-98.7 to 25.0] | -39.4 [-107.6 to 28.8]

10. Secondary Outcome: Change in Event-based Claudication Index
Description: Event-based claudication index (ratio of walking events to upright events) participants undertake in a day.
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: calculated ratio index
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
calculated ratio index
  Change from baseline to end of intervention (6 weeks) | -0.4 [-1.2 to 0.3] | -0.4 [-1.1 to 0.3] | 0.9 [-1.0 to 2.7] | -0.2 [-1.1 to 0.7]
  Change from baseline to follow-up (18 weeks) | -1.2 [-2.5 to 0.1] | -0.7 [-3.2 to 1.7] | 0.0 [-1.0 to 1.0] | -0.6 [-1.0 to -0.2]

11. Secondary Outcome: Intermittent Claudication Questionnaire (ICQ)
Description: Disease specific quality of life questionnaire. ICQ scores range from 0 to 100, with lower scores representing better health status and less impact of claudication
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Change from baseline to end of intervention (6 weeks) | 4.5 [-1.3 to 10.2] | 5.6 [0.3 to 10.8] | 8.5 [1.7 to 15.3] | 9.6 [3.5 to 15.7]
  Change from baseline to follow-up (18 weeks) | 4.4 [-0.4 to 9.2] | 2.3 [-3.9 to 8.5] | 9.3 [1.9 to 16.8] | 8.0 [3.2 to 12.7]

12. Secondary Outcome: Short-Form 36 Questionnaire- Physical Component
Description: Generic quality of life questionnaire, physical domain. The SF-36 Physical Component Summary (PCS) ranges from 0-100, with higher scores representing better outcomes.
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Change from baseline to end of intervention (6 weeks) | 1.4 [-1.4 to 4.3] | 0.0 [-3.3 to 3.3] | -5.2 [-8.5 to -1.8] | -4.5 [-8.4 to -0.7]
  Change from baseline to follow-up (18 weeks) | -0.6 [-3.4 to 2.2] | 1.0 [-2.6 to 4.6] | -3.7 [-5.5 to -1.8] | -3.3 [-7.2 to 0.7]

13. Secondary Outcome: McGill Pain Questionnaire (MPQ) Pain Rating Index (PRI)
Description: Pain quality questionnaire. The MPQ-PRI ranges from 0-78, with lower scores representing less pain and higher scores representing worse pain.
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Change from baseline to end of intervention (6 weeks) | 4.3 [-0.8 to 9.5] | 3.5 [-4.0 to 11.1] | -5.9 [-9.9 to -1.9] | -6.5 [-12.3 to -0.6]
  Change from baseline to follow-up (18 weeks) | 2.5 [-1.3 to 6.3] | 2.6 [-2.4 to 7.6] | -7.4 [-11.0 to -3.8] | -3.0 [-8.1 to 2.1]

14. Secondary Outcome: Visual Analogue Scale (VAS)
Description: Average Pain intensity in the past 7 days. The average pain intensity VAS ranges from 0-100 mm, with lower scores indicating less pain and better outcomes.
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Change from baseline to end of intervention (6 weeks) | -0.7 [-2.2 to 0.8] | -1.0 [-2.4 to 0.3] | -2.0 [-3.3 to -0.7] | -1.5 [-3.1 to 0.0]
  Change from baseline to follow-up (18 weeks) | -1.2 [-2.7 to 0.2] | -1.4 [-3.4 to 0.6] | -1.8 [-3.1 to -0.4] | 0.1 [-1.4 to 1.6]

15. Secondary Outcome: Brief Illness Perception Questionnaire (IPQ)
Description: The Brief IPQ uses 0-10 scales. Higher scores indicate worse perceptions (greater perceived consequences, concern, emotional impact, chronicity).
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Change from baseline to end of intervention (6 weeks) | -1.7 [-6.8 to 3.5] | 0.6 [-5.0 to 6.3] | -7.7 [-12.8 to -2.5] | -8.1 [-15.1 to -1.0]
  Change from baseline to follow-up (18 weeks) | -1.5 [-6.2 to 3.1] | 1.0 [-5.3 to 7.3] | -3.2 [-8.9 to 2.4] | -5.6 [-10.9 to -0.3]

16. Secondary Outcome: Geriatric Depression Scale (Short Form) (GDS-SF)
Description: Depression questionnaire. The GDS-SF ranges 0-15, with higher scores reflecting more depressive symptoms.
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Change from baseline to end of intervention (6 weeks) | -1.5 [-3.3 to 0.2] | -0.8 [-3.5 to 2.0] | -1.8 [-4.0 to 0.3] | -1.2 [-2.6 to 0.2]
  Change from baseline to follow-up (18 weeks) | -0.9 [-3.2 to 1.3] | 0.2 [-2.8 to 3.2] | -2.2 [-4.8 to 0.4] | -1.0 [-2.3 to 0.3]

17. Secondary Outcome: Pain Self-Efficacy Questionnaire (PSEQ)
Description: The PSEQ total score ranges from 0-60, with higher scores indicating better pain self-efficacy and more positive outcomes.
Time Frame: Baseline, 6 weeks (post-intervention), 18 weeks (follow-up)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Change from baseline to end of intervention (6 weeks) | 1.0 [-4.2 to 6.2] | 0.8 [-2.5 to 4.2] | 5.2 [-1.5 to 11.8] | 6.9 [1.7 to 12.1]
  Change from baseline to follow-up (18 weeks) | 1.9 [-3.7 to 7.6] | 0.4 [-5.5 to 6.3] | 5.8 [-1.8 to 13.4] | 3.6 [-1.9 to 9.1]

18. Secondary Outcome: SF-36 Mental Component Score
Description: SF-36 Quality of life scale - mental component. The SF-36 MCS ranges 0-100 (or norm-based mean 50, SD 10), with higher scores representing better outcomes.
Time Frame: Baseline, end of intervention and follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education and Placebo TENS | Patient-Centred Education + Active TENS
Number analyzed (Participants) | 14 | 14 | 14 | 14
units on a scale
  Change from baseline to end of intervention (6 weeks) | -2.8 [-7.6 to 2.0] | 0.5 [-5.9 to 7.0] | -3.0 [-9.4 to 3.4] | -1.8 [-6.8 to 3.2]
  Change from baseline to follow-up (18 weeks) | -0.1 [-4.4 to 4.3] | 0.1 [-7.8 to 8.0] | -2.7 [-7.2 to 1.7] | -0.4 [-4.7 to 4.0]

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Active TENS: Active TENS group
- Placebo TENS: Placebo TENS group
- Patient-Centred Education + Active TENS: Patient-Centred Education + Active TENS group
- Patient-Centred Education: Patient-Centred Education group
Arm/Group | Active TENS | Placebo TENS | Patient-Centred Education + Active TENS | Patient-Centred Education
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14 | 1/14 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TENS (N=14) | Placebo TENS (N=14) | Patient-Centred Education + Active TENS (N=14) | Patient-Centred Education (N=14)
Itching on leg due to TENS electrodes (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Three minor adverse events were reported throughout the study, all relating to a slight itching reaction to the TENS electrodes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03204825/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT03204825/SAP_001.pdf